## Informed Consent

PROJECT: THE USE OF LAVENDER ESSENTIAL OIL OR COLOSTRUM AS ADJUNCTIVE ANALGESIA TO SUBLINGUAL FRENOTOMY ON HEALTHY TERM NEONATES

| I, (name and surname)(father/mother/legal guardian of patient) |
|---|
| - I have read the information sheet provided to me |
| - I have been clearly informed of the purpose of the research and have received sufficient information |
| - I have spoken to (name of investigator) |
| - I have been able to ask questions about the study and I have been informed that any other questions related to the study will be answered by e-mail in a timely manner. |
| - I understand that participation is voluntary |
| - I understand that I can stop participating in the study whenever I want, and without having to give explanations |
| - I have been informed that the data from this research are strictly confidential and will not be used for any other purpose outside the study without consent |
| - I have been informed that my child's personal data will be protected according to the Organic Law 3/2018, of December 5, 2018, on the Protection of Personal Data and Guarantee of Digital Rights, and will be used only for purposes specified in the information sheet |
| - I understand that I have the right to access, rectification, cancellation and opposition of my child's personal data as provided by the Organic Law 3/2018 of December 5, 2018, on the Protection of Personal Data and Guarantee of Digital Rights |
| - I have been informed that I may receive information about the results of the study and I give my consent for the participation of my child in the study, as well as access to my child's data under the conditions detailed in the information sheet |
| - I understand that a signed copy of this informed consent will be given to me |
| Parents (both) |
| In the event that only one parent authorizes, the authorizing parent must state one of the following: |
| ☐ I confirm that the other parent does not object to our child's participation in the study participation |
| ☐ The undersigned is the sole legal guardian |
| Signature of the participant's parent Signature of the investigator |